CLINICAL TRIAL: NCT03228121
Title: Crossover Blinded Trial of Cell Therapy Versus Placebo in COPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment did not meet expectations
Sponsor: Lung Institute (Industry)
Responsible Party: Principal Investigator, Melissa Rubio, PhD, APRN, Principal Investigator, Lung Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LI003
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: COPD; Emphysema or COPD; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: 0 participants will be recruited for each arm of the study.
  Cohort A will receive three days of cell therapy using the venous procedure (three consecutive days of blood harvest, cell separation and cell application). Cohort A will return in three months and receive three consecutive days of placebo.
  Cohort B will receive three consecutive days of placebo. Cohort B will return in three months and receive three consecutive days of cell therapy using the venous procedure.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the on-site PI and research nurse administering the treatment or placebo will know which group the participant belongs to. Patients are blinded. All follow-up contact and measurement of outcomes will be done by off-site research nurses who are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Cohort A (Treatment Then Placebo group) will receive three days of cell therapy using the venous procedure (three consecutive days of blood harvest, cell separation and cell application). Cohort A will return in three months and receive three consecutive days of placebo.
  Interventions: Procedure: Treatment Then Placebo
- Cohort B (Experimental): Cohort B (Placebo Then Treatment group) will receive three consecutive days of placebo. Cohort B will return in three months and receive three consecutive days of cell therapy using the venous procedure.
  Interventions: Procedure: Placebo Then Treatment

INTERVENTIONS:
Procedure: Treatment Then Placebo — Cohort A will receive stem cells/PRP infusion during round one then placebo of normal saline infusion during round two.
  Arms: Cohort A
Procedure: Placebo Then Treatment — Cohort B will receive placebo of normal saline infusion during round one then stem cells/PRP infusion during round two.
  Arms: Cohort B

SUMMARY:
The aim of this randomized, controlled crossover designed study is to compare the outcomes of receiving autologous, adult stem cells versus placebo among participants with chronic obstructive pulmonary disease (COPD). The study is limited to self-funded participants with a diagnosis of COPD. The study, along with others at the Lung Institute, have received full review and approval of an Institutional Review Board.

DETAILED DESCRIPTION:
The purpose of the Lung Institute is to collect, minimally process, and administer a person's own stem cells and/or platelet rich plasma and deliver the product back to the patient same-day through an intravenous catheter. This study is limited to patients diagnosed with chronic obstructive pulmonary disease (COPD) and is a double-blinded prospective, cohort trial using cross-over methodology. The aim of this study is to determine if stem cell therapy is better than placebo among a group of patients with COPD.

50 participants will be recruited for each arm of the study.

Cohort A will receive three days of cell therapy using the venous procedure (three consecutive days of blood harvest, cell separation and cell application). Cohort A will return in three months and receive three consecutive days of placebo.

Cohort B will receive three consecutive days of placebo. Cohort B will return in three months and receive three consecutive days of cell therapy using the venous procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients are included in treatment by self-referral and after consultation with a designated patient coordinator who determines initial eligibility, and then by the clinic nurse practitioner or physician of Lung Institute who determines final eligibility for inclusion. Patients must be diagnosed with chronic obstructive pulmonary disease (COPD) and be able to travel to the Dallas clinic location.

Exclusion Criteria:

* Patients who are unable to provide informed consent, pregnant patients, prisoners, non-English speakers, patients with a history of cancer within the past 5 years, patients with active tuberculosis or pneumonia. Patients without a documented COPD diagnosis are excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life Score | 3 months, 6 months following each treatment
  Change in QOL score from baseline to 3 months and 6 months following each treatment

SECONDARY OUTCOMES:
Change in FEV1 | 6 months following each treatment
  Change in FEV1 from baseline to 6 months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Lung Institute Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No